CLINICAL TRIAL: NCT03964636
Title: Contraceptive Pills and Retinal Vascularization (Piluret)
Brief Title: Contraceptive Pills and Retinal Vascularization
Acronym: PILURET
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: VVR_2019_6
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Combined Oral Contraceptives Intake
Keywords: OCT-A; combined oral contraceptives
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- no contraceptive intake
  Interventions: Diagnostic Test: OCT-A (optical coherence tomography)
- combined 1st/2nd generation oral contraceptives intake
  Interventions: Diagnostic Test: OCT-A (optical coherence tomography)
- 3rd/4th generation combined oral contraceptives intake
  Interventions: Diagnostic Test: OCT-A (optical coherence tomography)

INTERVENTIONS:
Diagnostic Test: OCT-A (optical coherence tomography) — Included patients will have an OCT-A and will be questioned about their medical and ophthalmologic history, and their oestro-progestative contraceptive intake.

SUMMARY:
The main hypothesis is the taking of combined 1st and 2nd generation or 3rd and 4th generation oral contraceptives is associated with a change in retinal micro-vascularization compared to the absence of combined oral contraceptive intake.

Women of childbearing age will be recruited during their ophthalmologic consultation at the Rothschild Foundation, an OCT-A will be realized and data relating to their medical and ophthalmologic history and their oestro-progestative contraceptive intake will be collected.

The objective is to find an association between retinal vascular density and combined oral contraceptives intake.

ELIGIBILITY:
Inclusion criteria

* for the control group : No Estro-progestin contraceptive treatment (oral, transdermal) for at least 6 months
* for the cases under combined 1st and 2nd generation pills : Estro-progestin contraceptive treatment for at least 6 months
* for the cases under combined 3rd and 2th generation pills: Estro-progestin contraceptive treatment for at least 6 months

Exclusion criteria:

* Menopausal woman
* Ametropia greater than + 3 hyperopia diopters or-3 myopia diopters
* Astigmatism greater than 2 dioptres
* Smoking patient (cigarette or e-cigarette)
* Caffeine intake within 2 hours prior to the OCT-A exam
* Any known retinal pathology
* Antecedent of deep vein thrombosis or deep arterial thrombosis

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women of chilbearing age presenting to an ophthalmologic consultation at the Foundation Rothschild will be included in one of the 3 groups: no contraceptive intake, combined 1st/2nd generation oral contraceptives and 3rd/4th generation combined oral contraceptives, if they meet the inclusion and non-inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Density of retinal vascular Plexus (quantitative variable expressed as a percentage) using OCT-A. | At the inclusion consultation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No